CLINICAL TRIAL: NCT06284343
Title: Development and Validation of a Risk Prediction Model for Venous Thromboembolism in Gynecological Cancer Patients Undergoing Systemic Antineoplastic Treatment: The Gynecological Cancer Associated Thrombosis (GynCAT) Study
Brief Title: The Gynecological Cancer Associated Thrombosis (GynCAT) Study
Acronym: GynCAT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Fondazione Umberto Veronesi (Other)
Responsible Party: Principal Investigator, Pola Roberto, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6414
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer-associated Thrombosis; Venous Thromboembolism; Gynecologic Cancer; Ovarian Cancer; Cervix Cancer; Endometrial Cancer; Vaginal Cancer
Keywords: Thrombosis; Venous thromboembolism; Cancer; Ovarian Cancer; Vaginal Cancer; Endometrial Cancer; Gynecologic Cancer
MeSH Terms: conditions — Venous Thromboembolism; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Thrombosis; Neoplasms | interventions — Anticoagulants; Heparin, Low-Molecular-Weight; apixaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by Gynecologic Cancer undergoing systemic antineoplastic treatment: Study population will consist of subsequent patients prospectively enrolled at the time of prescription of a new line of systemic antineoplastic treatment for a gynecologic oncological disease, defined as ovarian, tubal, uterine, cervical, vaginal, or vulvar neoplasm
  Interventions: Drug: Anticoagulant

INTERVENTIONS:
Drug: Anticoagulant — Prescription of pharmacological thromboprophylaxis according to current clinical practice and international guidelines recommendation
  Other Names: Low Molecular Weight Heparin; Apixaban; Rivaroxaban

SUMMARY:
GynCAT is a prospective cohort study that will be conducted on female patients with gynecologic malignancies scheduled for systemic antineoplastic treatment, aiming at development and validation of a Risk Assessment Model (RAM) for Venous Thromboembolism (VTE) in this specific population.

DETAILED DESCRIPTION:
Cancer patients are burdened by an increased risk of venous thromboembolism (VTE), which has a significant impact on morbidity and mortality. Existing Risk Prediction Models (RPMs), including the widely accepted Khorana Risk Score (KRS), have some limitations when used in certain tumor site populations, such as gynecological cancers. Notably, gynecological patients exhibit a variable risk of VTE based on their specific tumor sites, with ovarian cancer representing the highest risk. Moreover, currently available RPMs lack validation in a broad gynecological population and may fail to effectively stratify VTE risk.

GynCAT is a prospective cohort study that will be conducted on female patients with gynecologic malignancies scheduled for systemic antineoplastic treatment. During the screening phase, symptomatic VTE will be excluded, and KRS will be assessed. Pharmacological thromboprophylaxis will be considered and prescribed at clinical judgement, for patients with a KRS score of 3 or higher. Clinical, hematological, biochemical, coagulation, and genetic variables will be collected. Follow-up will last for the entire duration of the antineoplastic treatment line, and VTE events, bleeding events, and mortality will be recorded.

The primary objective is the development and validation of an RPM for VTE in gynecologic cancer patients undergoing systemic antineoplastic treatment. Secondary objectives are evaluation of the predictive value of the identified model, comparing it with existing general oncology RPMs; assessment of its performance in predicting mortality; evaluation of VTE incidence in patients with KRS≥3 receiving thromboprophylaxis; identification of risk factors for bleeding in this patient population.

The sample size calculation is based on an estimated VTE incidence of 5% over a mean follow-up of 12 months. Hence, a sample size of at least 1,200 patients in the derivation cohort is considered sufficient for the determination of a risk prediction model incorporating up to six predictor variables. A split-sample method will be used, with two-thirds of the study participants randomly assigned to the model derivation cohort (n=1,200) and one-third (n=600) to an independent validation cohort. The total number of patients recruited in the study will thus be of 1,800. A competing risk survival analysis with Fine & Gray model will be used to study the association between prognostic variables and VTE occurrence, considering death as a competitive risk. The RPM will be identified through a bootstrap approach to reduce the risk of overfitting. Discrimination power of the RPM will be assessed using time-dependent Receiving Operating Characteristic curve, and model calibration will be evaluated graphically and with the calculation of relative calibration slopes.

In conclusion, this prospective cohort study aims to overcome the limitations of current RPMs in gynecologic cancer patients, improving the accuracy of VTE risk stratification in this population.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Diagnosis of gynecologic neoplasm (ovarian, tubal, uterine, cervical, vaginal, vulvar neoplasm);
* Planned new line of systemic antineoplastic treatment;
* Age of 18 years or older;
* Accordance of Informed Consent.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Indication to receive therapeutic dose anticoagulant therapy (e.g., atrial fibrillation, mechanical heart valve);
* Diagnosis of symptomatic VTE at the time of screening for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients affected by Gynecologic Cancer
Study Population: Study population will consist of subsequent patients prospectively enrolled at the time of prescription of a new line of systemic antineoplastic treatment for a gynecologic oncological disease, defined as ovarian, tubal, uterine, cervical, vaginal, or vulvar neoplasm.
  Patients will be recruited in the setting of the Gynecologic Oncology Day Hospital and evaluated by the Thrombosis Clinic of the Agostino Gemelli University Polyclinic Foundation I.R.C.C.S. in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Venous thromboembolism | Follow-up will continue until one of the following censoring events will occur: • EpPatients will be evaluated with one in-person medical visit at enrollment, followed by one telephone visit and one in-person examination at 6 and 12 months, respectively.
  Venous Thromboembolism (VTE) diagnosis will be assigned in case of objective confirmation by venous duplex ultrasonography and/or contrast enhanced CT and/or MRI and/or ventilation/perfusion SPECT.
  In case of death during follow-up, clinical documentation and/or autopsy findings, if available, will be reviewed to assess for the presence of a possible diagnosis of fatal pulmonary embolism.
  VTE events will be independently judged by an external committee, constituted by Angiology and Radiology experts, blinded to patients' clinical history and laboratory parameters. Incidentally detected VTE events will be considered as events, provided their eligibility by the aforementioned external committee.

SECONDARY OUTCOMES:
Number of Participants with Bleeding events (major and clinically relevant non-major bleeding) | Follow-up will continue until one of the following censoring events will occur: • EpPatients will be evaluated with one in-person medical visit at enrollment, followed by one telephone visit and one in-person examination at 6 and 12 months, respectively.
  After acquisition and review of the clinical documentation related to a hemorrhagic event, bleeding will be assigned if requirements for major or clinically relevant nonmajor bleeding are met, as defined by the International Society on Thrombosis and Haemostasis (ISTH)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pola, PhD; MD, Principal Investigator — Agostino Gemelli University Polyclinic Foundation IRCCS; Paolo Santini, MD, Study Chair — Agostino Gemelli University Polyclinic Foundation IRCCS
Locations (1):
- Agostino Gemelli University Polyclinic Foundation IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided